CLINICAL TRIAL: NCT02077257
Title: A 12-Week, Randomized, Open-Label, Multicenter Study Exploring Low-Density Lipoprotein Cholesterol Lowering Efficacy and Safety of Rosuvastatin 20 mg/Day Compared to10 mg/Day in Chinese Patients With Acute Coronary Syndromes
Brief Title: LDL-C Lowering Efficacy and Safety of Rosuvastatin 20 mg/Day to10 mg/Day in Chinese ACS(Acute Coronary Syndrome) Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Committee of Cardio-Cerebral-Vascular Diseases of GSC (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSE
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin 20mg (Other): Rosuvastatin 20 mg/d
  Interventions: Drug: Rosuvastatin
- Rosuvastatin 10mg (Other): Rosuvastatin 10 mg/d
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20 mg/d compared to 10 mg/day

SUMMARY:
This is a 12-week, randomized, open-label,,multicenter, Phase IV study exploring LDL-C lowering efficacy of Rosuvastatin 20 mg/d compared to 10 mg/day Chinese ACS patients.The Randomized Treatment Period is preceded by a 24hours Screening Period. The study flow chart (Figure 1) depicts the 2 periods which comprise the study. These periods are described as follows:

1. Screening Period (Day -1 through Day 1) This period consists of Visits 1 and 2. Subjects entering the Screening Period are required to meet the inclusion criteria. All subjects will be instructed to follow the current TLC(therapeutic lifestyle change)dietary guidelines for the duration of the trial.
2. 12-week Randomized Treatment Period (Day 1 through Week 12) This period consists of Visits 2, 3, 4, and 5. Eligible subjects will be randomized at Visit 2 to each treatment group: Rosuvastatin 20 mg orRosuvastatin10 mg. Treatment will be administered once daily for 12 weeks.

A total of 450valid subjects in each of the Rosuvastatin arms are required, in order to test the hypothesis of superiority for comparison of LDL-C levels between Rosuvastatin20 mg and Rosuvastatin10 mg(see Section 6.1 for more details).

The Study visit schedule(Table 2) indicates the number and timing of the planned visits. The visit schedule must be within time window. At the final visit, it is the responsibility of the investigator to ensure the subject is offered an selected appropriate type of lipid-lowering therapy.

Scheduled Visit3,4,5 will have a visit window of ±2 days. Subjects who attend a clinic visit without fasting (at least 12 hours) should be asked to return within 2 days for another clinic visit after fasting for at least 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year old males and non-child-bearing period females.
* Clinical diagnosed with acute coronary syndrome including NSTE-ACS ,MI and STEMI.
* Patients with STEMI((ST segment elevation myocardial infarction) and NSTEMI(non-ST segment elevation myocardial infarction) will be recruited within 48 hours of symptom onset.
* The LDL-C≥70mg/dL one week before randomization.
* The TG<500mg/dL one week before randomization.
* No cholesterol-lowering drugs (including lipid lowering dietary supplements, antioxidants, or food additives) during 4 weeks before randomization.
* Sign the ICF(inform consent form)

Exclusion Criteria:

* Acute pulmonary edema, severe congestive heart failure,
* acute moderate mitral regurgitation, acute ventricular septal perforation,
* severe arrhythmia (ventricular fibrillation, sustained ventricular tachycardia, complete heart block), sepsis, acute pericarditis,
* any evidence of systemic or pulmonary embolus within the preceding 4 weeks.
* Coronary artery bypass graft within the preceding 3 months; percutaneous coronary intervention within the preceding 6 months.
* A history of hypersensitivity of statins and other severe complication.
* child-bearing women
* hypothyroidism,
* active liver disease or dysfunction including agnogenic serum transaminase sustained elevation or higher than 3 times ULN(upper limit of normal)
* severe anemia (hemoglobin,hematocrit < 28%),
* Patients with myopathy or serum creatine kinase > 3 times the upper limit of normal not caused by myocardial injury.
* A history of psychiatric disorders
* A history of jejunoileal bypass or gastric bypass surgery
* Currently take steroids therapy
* Currently take phenytoin sodium,phenobarbital,carbamazepine (which may primary efficacy endpoint)
* Diagnosed with malignant within 5 years
* Severe renal function damage (creatinine clearance rate<30 ml/min)
* Concurrent use ciclosporin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
LDL-C absolute value and percent change from baseline | 12 weeks
  Rosuvastatin 20mg/d ( absolute value and percent change from baseline) compared with that of Rosuvastatin 10mg/d (absolute value and percent change from baseline) in lowering LDL-C averaged over measurements at 12 weeks.

SECONDARY OUTCOMES:
blood lipid goal achievement rate(LDL-C <70 mg/dl or 50% reduction) | 6 week
  Efficacy of Rosuvastatin 20 mg/d vs Rosuvastatin 10 mg/don blood lipid goal achievement rate(LDL-C <70 mg/dl or 50% reduction) at Weeks 6
blood lipid goal achievement rate(LDL-C <70 mg/dl or 50% reduction) | 12 weeks
  Efficacy of Rosuvastatin 20 mg/d vs Rosuvastatin 10 mg/don blood lipid goal achievement rate(LDL-C <70 mg/dl or 50% reduction) at Weeks 12
Percent change from baseline in TC,HDL-C, TG, nonHDL-C (non HDL-C = [TC-HDL-C]), ApoA-I, ApoB, LDL-C/HDL-C, TC/HDL-C, non HDL-C/HDL-C, ApoB/ApoA-I and LDL-C | 6weeks
  Percent change from baseline in TC(total cholesterol), HDL-C(high density lipid cholesterol), TG(triglyceride), nonHDL-C (non HDL-C = [TC-HDL-C]), ApoA-I(apolipoprotein A ), ApoB(apolipoprotein B ), LDL-C/HDL-C, TC/HDL-C, non HDL-C/HDL-C, ApoB/ApoA-I and LDL-C at Weeks 6 .
Percent change from baseline in TC, HDL-C, TG, nonHDL-C (non HDL-C = [TC-HDL-C]), ApoA-I, ApoB, LDL-C/HDL-C, TC/HDL-C, non HDL-C/HDL-C, ApoB/ApoA-I and LDL-C | 12 weeks
  Percent change from baseline in TC, HDL-C, TG, nonHDL-C (non HDL-C = [TC-HDL-C]), ApoA-I, ApoB, LDL-C/HDL-C, TC/HDL-C, non HDL-C/HDL-C, ApoB/ApoA-I and LDL-C at week 12
Percent change from baseline in the level of hsCRP(high-sensitivity C-reactive protein), an inflammatory marker | 6 weeks
  Percent change from baseline in the level of hsCRP, an inflammatory marker, following 6 weeks
Percent change from baseline in the level of hsCRP, an inflammatory marker, | 12 weeks
  Percent change from baseline in the level of hsCRP, an inflammatory marker, following 12 weeks
incidence and severity of adverse events | 12 weeks
abnormal physical examination findings | 12 weeks
abnormal laboratory values | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dayi Hu, Doctor, Principal Investigator — Beijing university People's hospital; Changsheng Ma, Doctor, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China